CLINICAL TRIAL: NCT04785911
Title: Use of the Modified PUQE ( Pregnancy -Unique Quantification of Emesis ) Score on Admitted Cases of Hyperemesis Gravidarum (HG) to Guide Response to Treatment
Brief Title: Use of the Modified PUQE Score on Admitted Cases of Hyperemesis Gravidarum (HG) to Guide Response to Treatment
Status: Completed | Type: Observational
Sponsor: Tasnem Abo-elouon (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Tasnem Abo-elouon, Principal investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: 17101318
Record Dates: First submitted 2021-01-21; First posted 2021-03-08 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Hyperemesis Gravidarum
Keywords: PUQE score
MeSH Terms: conditions — Hyperemesis Gravidarum | interventions — Steroids; Histamine Antagonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Antiemetic Combinations — Evaluation of response to treatment of hyperemisis gravidarum (antiemetics and other methods ) by PUQE score
  Other Names: Steroids; Anti histamine

SUMMARY:
Use of the PUQE score to judge the need for admission in cases of hyperemesis gravidarum Evaluation of the response to treatment by the PUQE score

DETAILED DESCRIPTION:
Nausea and nomiting of Pregnancy (NVP) affects up to 80% of pregnant women . Severe NVP is one of the most common indications for hospital admission among pregnant women, with typical stays of between 3 and 4 days . Onset of NVP is in the first trimester. It typically starts between the fourth and seventh weeks of gestation, peaks in approximately the ninth week and resolves by the 20th week in 90% of women. If the initial onset is after 10+6 weeks of gestation, other causes need to be considered There is a broad spectrum of nausea and vomiting of pregnancy (NVP) severity, ranging from mild, occasional nausea to severe, intractable vomiting requiring hospitalisation (hyperemesis gravidarum). Hyperemesis gravidarum(HG) is defined severe, protracted nausea and vomiting associated with weight loss of more than 5% of prepregnancy weight, dehydration and electrolyte imbalances. The exact underlying pathophysiology is unknown, but etiology is believed to be multifactorial, including endocrine, gastrointestinal and environmental factors.5 Risk factors include lower maternal age, primigravidity, lower socioeconomic background and non-smoking status.

Admission for hyperemesis gravidarum depends on clinical impression by the attending or referring physician. There is a need for classification the severity of NVP to restrict admission to those who need admission. An objective and validated index of nausea and vomiting such as the Pregnancy-Unique Quantification of Emesis (PUQE) score may be used for this purpose.

This questionnaire contains three questions regarding the time-span of nausea, vomiting and retching respectively, as well as one question assessing the global psychological and physical quality of life (QOL). Initially the questionnaire evaluated symptoms during last 12 hours, but it has been modified to encompass 24 hours as well as the whole of first trimester of pregnancy The PUQE questionnaire was used in several studies to assess the effect of antiemetic treatments for emesis and hyperemesis . In this study, the role of PUQE in evaluating need for inpatient admission will be studied. Also, the response to treatment inside the hospital will be assessed

ELIGIBILITY:
Inclusion Criteria:

* women hospitalized due to hyperemesis gravidarum with at least two out of three criteria; dehydration, weight loss > 5% of prepregnancy weight (if known) or electrolyte imbalance/ketonuria.
* Gestational age between 6_16 weeks.

Exclusion Criteria:

1. Women Suffered from other diseases causing nausea and vomiting :

   * gastritis
   * renal diseases
   * Hepatic disorders
   * Throid disorders
2. the gestational length was more than 16 weeks at inclusion.

Ages: 16 Years to 46 Years | Sex: Female
Age Groups: Child, Adult
Study Population: All admitted pregenent cases complaining of hyperemisis gravidarum
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-09-05 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Detect improvement of patients by 1- daily scor of PUQE score 2-BMI by kg/m2 change from day of admission to day of discharge | Basline
  We can assess severity and change by daily score which detected by daily PUQE score and pre gestational BMI by kg/m2 and BMI by kg/m2 of pregenent women with hyperemisis from day of admission to hospital to day of discharge To descripe the PUQE score full text with scoring range will be attached Total score is sum of replies to each of the three questions. PUQE-24 score: Mild ≤ 6; Moderate = 7-12; Severe = 13-15.
  Motherisk PUQE-24 scoring system
  1. the last 24 hours, for how long have you Felt nauseated or sick to your stomach? Not at all (1 ) 1hour or less (2) 2-3 hours(3) 4-6 hours (4) More than 6 hours (5)
  2. In the last 24 hours have you vomited Or thrown up? 7 or more Times (5) 5-6 times (4) 3-4 times(3). 1-2 times(2) I did not throw up (1)
  3. In the last 24 hours how many times Have you had retching or dry heaves Without bringing anything up? No time (1) 1-2 times(2) 3-4 times(3) 5-6 times (4) 7 or more times (5)

CONTACTS AND LOCATIONS:
Locations (1):
- Tasnem iIbrahem Aboelouon, Asyut, Assuit, Egypt

REFERENCES:
- See also: Epidemiology of vomiting in early pregnancy. — http://europepmc.org/article/med/3903578